CLINICAL TRIAL: NCT04366037
Title: Effectiveness of Proprioceptive Exercises in Warm-up or Cool-down on Knee Injuries Prevention in Youthful Soccer Players.
Brief Title: Effectiveness of Proprioceptive Exercises in Soccer.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Ramón Jiménez Gómez del Pulgar, Physiotherapist, University of Alcala
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CEIM HU 2019-49
Record Dates: First submitted 2020-04-16; First posted 2020-04-28 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Knee Injuries
Keywords: proprioception; knee injuries; prevention; soccer; warm-up exercise; cool-down exercise
MeSH Terms: conditions — Knee Injuries | interventions — Warm-Up Exercise

STUDY DESIGN:
Intervention Model Description: Cuasiexperimental
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Experimental): This group performed their routine training
  Interventions: Other: Routine training
- Experimental 1 (Experimental): This group performed their routine training plus proprioceptive exercises in the warm-up.
  Interventions: Other: Routine training + proprioceptive exercise in warm-up
- Experimental 2 (Experimental): This group performed their routine training plus proprioceptive exercises in the cool-down
  Interventions: Other: Routine training + proprioceptive exercise in cool-down

INTERVENTIONS:
Other: Routine training — Training will be defined by each club coach
  Arms: Control group
Other: Routine training + proprioceptive exercise in warm-up — Training will be defined by each club coach, adding four proprioceptive exercises in warm-up:
  Exercise Description Duration Antero-posterior bipodal horizontal jump Players will jump forward and backward with both feet together, keeping their hands on their waists 30 seconds Unipodal lateral jump Players will perform single-leg lateral jump on both sides of a previously drawn line on the ground, and keeping their hands on their waists. 30 seconds per limb.
  Antero-posterior unipodal horizontal jump Players will jump forward and backward with one foot, keeping their hands on their waists 30 seconds per limb.
  Bipodal vertical jump with or whitout ball. Players will perform vertical jumps with both feet carrying a ball in their hands (this added difficulty will be optional). 30 seconds
  Arms: Experimental 1
Other: Routine training + proprioceptive exercise in cool-down — Training will be defined by each club coach, adding four proprioceptive exercises in cool-down:
  Exercise Description Duration Antero-posterior bipodal horizontal jump Players will jump forward and backward with both feet together, keeping their hands on their waists 30 seconds Unipodal lateral jump Players will perform single-leg lateral jump on both sides of a previously drawn line on the ground, and keeping their hands on their waists. 30 seconds per limb.
  Antero-posterior unipodal horizontal jump Players will jump forward and backward with one foot, keeping their hands on their waists 30 seconds per limb.
  Bipodal vertical jump with or whitout ball. Players will perform vertical jumps with both feet carrying a ball in their hands (this added difficulty will be optional). 30 seconds
  Arms: Experimental 2

SUMMARY:
SUMMARY Contextualization The knee is one of the joints that has more injuries reports in men's soccer. Nowadays there are different injury prevention protocols, but none of them specifically focus on the knee joint. Numerous studies have shown that proprioceptive work is more effective than traditional protocols.

Objective This study aims to test the effects of a proprioceptive exercise program included as part of warm-up or cool-down in preventing knee injuries and muscle performance in youth soccer players Methodology This is a quasi-experimental study with three intervention groups. One group will be control, another group will be experimental with the intervention in the warm-up phase, and another one experimental group with the intervention in the cool-down phase. The independent variable will be the proprioceptive exercises, the dependent variables will be the dynamic balance measured with the Y Balance Test, and the muscular performance measured with Counter Movement Jump and the 40m sprint. The confounding variables will be age, height, weight, and body mass index (BMI).

DETAILED DESCRIPTION:
Soccer is a high intensity sport, characterized by continuous changes of direction and high load unipodal actions, which generates high levels of stress in the lower limbs, particularly in the knees . Consequently, there is a high rate of lower limb injury in men's soccer, with the knee being one of the most frequent injured joint, with an average of 14% of injury records.

There are varied preventive strategies for this type of injury which are usually included in the warm-up. Popular protocols like FIFA 11+, HarmonKnee, Elis and Rosembaum, Prevent Injury and Enhance Performance Program, include strength exercises, stretching, balance and plyometry; and other protocols focus exclusively on plyometric exercises or strength exercises in soccer.

The results of these protocols usually show proprioception as one of the factors to be improved since it has been observed that it is a determining element in the prevention of injuries. Loss of proprioception has been shown to compromise motor and postural control.

Warm-up can benefit proprioception, stability and, thus, injury prevention. There are several recent studies showing that warm-up programs focused on proprioception are more successful at preventing injuries than traditional warm-ups in athletes.

On the other hand, current protocols, such as those proposed by the FIFA Medical and Research Center (F-MARC) and Hubscher, demand to study in a more isolated way which components of these programs are the most effective.

Another important feature of these programs is the time of training in which they are included. Although most of the studies consider more appropriate to carry them out as part of the warm-up, there is no consensus among the authors. Currently there is great controversy due to the lack of studies evaluating and comparing the effects of this type of program on key prevention parameters such as postural stability or lower limb strength as they are included before or after training. Studies that have analyzed the effects of performing preventive programs after training have shown similar gains in strength parameters, although the components of the program were mostly eccentric exercises.

However, to our knowledge, there are no studies so far comparing the effects of a preventive program based on postural stability exercises included before or after the main part of soccer training. For this reason, it is necessary to carry out a study that evaluates the effectiveness of a proprioceptive exercises program in the injurious incidence of the knee, postural stability and muscular performance of youth soccer players, comparing these effects according to the inclusion of this program as part of the warm-up or part of the cool-down of the training.

Objectives

1. -To compare the effects of a proprioceptive balance and force-explosive exercise program included in the warm-up phase or cool-down phase on the knee injuries incidence in youth soccer players.
2. -To assess the effects of a proprioceptive exercise program of balance and strength on the postural stability and muscular performance of youth soccer players.

METHODOLOGY Study design This quasi-experimental study was carried out with 3 intervention groups. The study will be carried out on soccer teams from the Community of Madrid. In each team there will be 3 intervention subgroups. Each team is divided into: a control group (CG), an experimental group in which the intervention will be performed in the warm-up phase (EG1) and an experimental group in which the intervention will be carried out in the coool-down phase. after the training or match (EG2). The CG will perform the training routine that the team used to do; the EG1 will execute the warm-up routine that the team normally do plus the balance exercises of the HarmoKnee program; and the EG2 will do the warm-up routine they used to do at the training or game, plus, to finish, perform the balance exercises of the Harmoknee program to cool-down.

Randomization will be stratified depending on the soccer club, guaranteeing the blinding of the assignment sequence by the distribution of opaque or sealed letters. Study will start on preseason, that take place on January 2020. Randomization and intervention will be carried out in each club's soccer pitch. The exposition dedicated to the importance of training proprioception at injury prevention and muscular performance to the primarily responsable doctors and sport managers as the measurement taking to the players will be done the first day of the team training. The same day, the multi-modal, HarmoKnee based-on balance exercises that the experimental groups must do will be shown and taught. Intervention will last 8 weeks. Physiotherapists will examine the execution of the exercises corresponding to each program in each training day or match to be able to make corrections if necessary and assure the compliance to the injury prevention program. Measurements will be taken after the intervention and a 1-month after the intervention a third and last measurement will be done. The measurements the physiotherapists will take are: age, weight, height, body mass index (BMI). Additionally, players will take these following tests, which will be taken before, after, and one month after the intervention: Y balance Test, Counter Movement Jump and 40-m Sprint Performance. Since the beginning of the intervention (January 2020) until the past 3 months a weekly register of the number of knee injuries that will be written in a Word document and will be verified in person by the investigators and the medical service of the team. Any missing time of training or any physical complaint (with no need of medical assistance) by a player that comes of a match/ training will be considered as an injury.

The consensus found in the medical literature to classify the injury gravity - and the most used criteria for it in similar studies to this (it is time-based: (on number of days) from the moment that the injury occurs to the day that the player is able to fully return to training and playing matches. The classification is described on the next table (Table 1):

TABLE 1. INJURY CLASSIFICATION DEFINITION INJURY DURATION Slight discomfort 0 days Minimum injury 1-3 days Mild injury 4-7 days Moderate injury 8-28 days Severe injury < 28 days Injuries that cause the end of the sportive career

Participants Sample size calculation was estimated using GiPower 3.1.9.2., Windows version, using an ANOVA statistical test of repeated measures with an error α of 0,5, a potency of 0,95 for the 3 groups and 3 types of measurements with a result of 36 subjects, which effect size will be 0,7. Despite this, our objective will be to recruit a maximum of 60 subjects, that is to say, our sample will be comprehended between 36 and 60 subjects.

The recruitment will apply for soccer teams from Madrid Community. Ethical Aspects Before entering on the experimental phase, subjects will be informed of the intervention details. Revocation of study participation has been included in a final paragraph at the informed consent form. Study will be carried out following the Helsinki Declaration principles.

Obtained data will be confidential (by anonymity, a codification system and safekeeping). In addition, they will always be presented with due caution and guarantees, complying with the Organic Law 15/1999, of December 13th, on protection of personal data.

Codification procedure will be done by using the player's licence federation number, in a way of avoiding the manipulation of personal data. In the case where personal data manipulation will be needed, it will be the club coaches who provide that information, instead of being the investigators the ones who are in possession of that information.

Procedure:

Before starting the intervention, presidents, coaches, club's technical group, players and their parents (when needed) will be informed of the investigation project. For this purpose, investigators will make an exposition to the to the primarily responsable doctors and sport managers about the importance of injury prevention. Along the first session initial measurements and earlier mentioned tests will be taken. Plus, an information paper will be handed over the players , and another one for their parents and players of legal age along an informed consent form for the voluntary participation to the study (to the players plus, in the case they are minors, to theirs parents). Once informed consent form is signed by the players and their parents when needed, the measure register will begin.

Initial measures that will be used as confounding variables are: height (measured with a portable stadiometer SECA 217 in centimeters (cm)), weight (measured by a weight machine Tanita BC-545N in kilograms (kg)), BMI (the ratio of a person's weight (kg) to his or her height (m) squared), and age (years). Multimodal exercises are the independent variable. Dependent variables will be postural stability (Y Balance Test), lower limb strength (Counter Movement Jump) and speed (40 metre Sprint Performance). Tests will be taken after the teams have warmed-up.

Y balance test YBT is an instrument for functional evaluation for lower limb derived from Star Excursion Balance Test. To prepare this test, a "Y" letter is drawn on the ground with an adhesive band. The length on each of the three directions will be of 1,5 meters; there will be 90º between postero-medial axis (PMA) and postero-lateral axis (PLA); 135º between the PMA and anterior axis (AA) and 135º between AA and PLA . One of the lower limbs must be maintained in the convergence of those three directions and the other one must try to search for the anterior, postero-medial and postero-lateral Y directions. To do this test each individual must repeat 7 times the "Y", rest for 30 seconds between repetitions, and for limb changing, rest for a minute. 6 of 7 repetitions are for training and the measurement is taken on the seventh repetition. The execution of this test will be performed in unipodal standing, hands on waist, while the participant avoids loosing balance or stepping on the adhesive band with the "reaching" foot and keeps looking to an anterior direction . The measures to take will be: the distance the player has reached in each direction in centimeters, the length of the assessed lower limb (from anterior superior iliac spine to medial malleolus) in centimeters. After taking this measures the formula to be fulfilled will be: the result of the maximum distance the individual has reached divided by the length, multiplied by 100[(maximum distance in one of the directions/lower limb length) * 100]. This is the way to obtain the maximum length percentage. To accomplish reliable results, measures will be taken by 2 physiotherapists: each one will obtain the measures independently, to compare them afterwards, and obtain the IC of the test.

Counter movement jump CMJ is a vertical jump from a static and standing position. To execute the jump the individual must start from a 90º flex-extension position. The person being evaluated must place the hands on the hips, put his/her feet in a plantar flexion, and avoid to flex his/her knees or arching the back during the jump. The measurement will be done by using the mobile application MyJump2. The result is the height of the jump, measured in centimeters (cm).

40m sprint performance The players will make 2 maximum efforts of 40 metre sprint, resting 5 minutes between both sprints. It starts from a crouch position, with a hand contacting the ground. Both sprints will be evaluated with the mobile application MySprint . The result will be the speed in meters per second (m/s).

Once data is registered, randomization with opaque letters will start. Proprioceptive exercises program Proprioception exercises will be the next: antero-posterior bipodal horizontal jump, unipodal lateral jump, antero-posterior unipodal horizontal jump and bipodal vertical jump with or without ball. The exercises will be repeted in two sets. The resting will always be of 2 minutes between exercises and 1 minute between sets of exercises. Exercises will be repeated three times a week (Tabla 2).

To select the exercises, authors have taken into account designs of programs done by previous studies.

TABLE 2. PROPRIOCEPTIVE EXERCISES PROGRAM

1. - Antero-posterior bipodal horizontal jump: Players will jump forward and backward with both feet together, keeping their hands on their waists for 30 seconds
2. - Unipodal lateral jump: Players will perform single-leg lateral jump on both sides of a previously drawn line on the ground, and keeping their hands on their waists for 30 seconds per limb.
3. - Antero-posterior unipodal horizontal jump: Players will jump forward and backward with one foot, keeping their hands on their waists for 30 seconds per limb.
4. - Bipodal vertical jump with or whitout ball: Players will perform vertical jumps with both feet carrying a ball in their hands (this added difficulty will be optional) for 30 seconds

Injury register Once a week, a knee injuries register will be written. It will be done by phoning the club's coach. Number of knee injuries will be registered in the ANNEX II Table. This register will record the number of new injuries that may occur each week, giving that number an absolute value. Also, it will differentiate between right or left leg.

The design section of the study gives the details about what is considered a knee injury in soccer.

Statistical analysis Data will be organized and analyzed with SPSS 18.00 version for Windows (IBM, Armonk, NY, EE.UU.). Statistical Significance level will be considered in a value of α= 0.05. In this study, according with the Saphiro Wilk test, in no case there won't be a number of subjects (n) higher or equal to 30 per group. Then, a normal contrast must be done. We will verify the normality of the main variables using the Shapiro-Wilk test. Plus, a descriptive analysis of the data will be done providing the mean +/- Standard Deviation (SD) of the normally distributed variables and median and interquartile ranges (Q1 and Q3) of the non-normally distributed varibles. Both independent variable and dependent variables are cuantitative. To establish intragroup comparatives of the three measurements (before intervention, after intervention, at week 8; and a 1 month post-intervention one): if the variable to manage is cuantitative and it adjusts to the normal distribution, ANOVA will be used on repeated measures, complemented with comparative tests by pairs of measures as Simple and Helmert contrasts. If the variable to manage is quantitative but doesn't adjust to normal distribution, ANOVA Friedman's test will be used, also complemented with comparative tests done by pairs of measures. To establish intergroup comparisons of each dependent variable: if dependent variable is normal, lineal regression or Pearson correlation coefficient will be used; if it is not normal, we will use Spearman's rank correlation coefficient or Kendall's Tau correlation coefficient. Variance homogeneity between groups will be studied using Levene's test for age, height, weight and BMI. To complete this analysis, effect size was calculated making use of Cohen's kappa coefficient (d) and confidence intervals at 95%.

ELIGIBILITY:
Inclusion Criteria:

* belong to a soccer club, belong to the category of men's youth soccer,
* Not having suffered any musculoskeletal injury to the lower limb during the previous 6 months to the start of the intervention

Exclusion Criteria:

* suffering a neurological condition,
* suffering severe hearing or visual conditions or performing proprioceptive exercises as part of the warm-up or calm down prior to the investigation

Ages: 16 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 36 (Estimated)
Dates: Start 2020-07-26 (Actual); Primary Completion 2020-08 (Estimated); Study Completion 2020-09 (Estimated)

PRIMARY OUTCOMES:
Y Balance Test | pre-intervention
  Dynamic balance has been tested using Y Balance Test
Y Balance Test | post-intervention
  Dynamic balance has been tested using Y Balance Test
Y Balance Test | 4 weeks post-intervention
  Dynamic balance has been tested using Y Balance Test

SECONDARY OUTCOMES:
counter movement jump | pre-intervention
  muscle performance has been tested using counter movement jump
counter movement jump | post-intervention
  muscle performance has been tested using counter movement jump
counter movement jump | 4 weeks post-intervention
  muscle performance has been tested using counter movement jump

OTHER OUTCOMES:
40-m sprint performance | pre-intervention
  muscle performance has been tested using 40-m sprint performance
40-m sprint performance | post-intervention
  muscle performance has been tested using 40-m sprint performance
40-m sprint performance | 4 weeks post-intervention
  muscle performance has been tested using 40-m sprint performance

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Romero-Franco, PhD, Study Director — University of the Balearic Islands
Locations (1):
- Universidad Alcala de Henares, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No